CLINICAL TRIAL: NCT06116760
Title: Anodal tDCS With Compensatory Audio-visual Training for Acquired Visual Field Defects After Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25C901
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Hemianopsia, Homonymous
Keywords: Homonymous Visual Field Defects; Hemianopia; Compensatory training; Audio-visual multisensory training; tDCS
MeSH Terms: conditions — Stroke; Hemianopsia

STUDY DESIGN:
Intervention Model Description: Three groups of participants were allocated to three different experimental treatments:
  Group 1: audio-visual training + ipsilesional occipital tDCS Group 2: audio-visual training + ipsilesional posterior parietal tDCS Group 3: audio-visual training + sham, placebo tDCS
Who Masked: Participant, Investigator
Masking Description: The tDCS device has a built-in function for double blind studies, i.e., the experimenters are not aware whether they are applying real or sham tDCS.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal Occipital tDCS + audio-visual training (Experimental): Anodal tDCS on ipsilesional occipital cortex. Anode electrode placed on O1/O2 (10-20 EEG system) and reference electrode placed on the contralateral forehead. Stimulation delivered at 2mA during the first 30 minutes of the audio-visual training.
  Interventions: Device: Anodal or sham tDCS; Behavioral: Audio-visual training
- Anodal Parietal tDCS + audio-visual training (Experimental): Anodal tDCS on ipsilesional posterior parietal cortex. Anode electrode placed on P3/P4 (10-20 EEG system) and reference electrode placed on the contralateral forehead. Stimulation delivered at 2mA during the first 30 minutes of the audio-visual training.
  Interventions: Device: Anodal or sham tDCS; Behavioral: Audio-visual training
- Sham tDCS + audio-visual training (Sham Comparator): Arm 3: sham tDCS. Half of participants with Group 1 montage, the other half with Group 2 montage. Stimulator is turned off after 30s of the audio-visual training.
  Interventions: Device: Anodal or sham tDCS; Behavioral: Audio-visual training

INTERVENTIONS:
Device: Anodal or sham tDCS — Anodal or sham tDCS (see "Arms") is applied during the execution of an audio-visual training.
Behavioral: Audio-visual training — 90 min/day x 10 days. Participants are seated in front of a 2 m × 2 m training board, at a distance of 1.2 m, in a dimly lit room. The board features 48 red light-emitting diodes (LED, diameter 1 cm, luminance 90 cd m2), distributed in six horizontal rows (eight lights per row). Forty-eight piezoelectric loudspeakers (0.4 W, 8Ω) are located above each light, producing a white-noise (80 dB, duration 100 ms).
  Spatio-temporally congruent, cross-modal, audio-visual stimuli are presented at one out of 48 possible positions on the board. Participants are instructed to look at the fixation point - at the center of the apparatus - and to move their eyes to detect the presence of the visual stimulus (duration=100 ms) by pressing right button of a wireless mouse.

SUMMARY:
Homonymous visual field defects (HVFDs) following acquired brain lesions affect independent living by hampering several activities of everyday life. Available treatments are intensive and week- or month-long. Transcranial Direct current stimulation (tDCS), a plasticity-modulating non-invasive technique, could be combined with behavioral trainings to boost their efficacy or reduce treatment duration. Some promising attempts have been made pairing occipital tDCS with visual restitution training, however less is knows about which area/network should be best stimulated in association with compensatory approaches, aimed at improving exploratory abilities, such as multisensory trainings.

In the present double-blind, sham-controlled study, we assess the efficacy of a multisensory training combined with tDCS. 3 groups of participants with chronic HVFDs underwent a 10-day (1.5 hrs/day) compensatory audio-visual training combined with either real anodal tDCS applied to the ipsilesional occipital tDCS (Group 1), or the ipsilesional posterior parietal cortex (Group 2), or a sham, placebo, tDCS (Group 3).

The training require the participants to orient their gaze training spatio-temporally congruent, cross-modal, audio-visual stimuli (starting from a central fixation) and press a button as quick as possible upon the detection of the visual stimulus. All stimuli are presented on 2mx2m panel embedded with 48 LEDs and loudspeakers (Bolognini et al., 2010, Brain Research)

All participants underwent a neuropsychological assessment of visuospatial functions prior to the beginning of the training (t0), at the end of the training (t1), and at 1-month (t2) and 4-month follow-up (t3). The assessment includes: a visual detection task, three visual search tasks (EF, Triangles, and Numbers; Bolognini et al., 2005, Brain), and a questionnaire about functional impact of the HVFDs in the activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

- Presence of chronic (>3 months) HVFD according to Neurophtalmological evaluation, due to acquired brain injury (i.e., stroke, traumatic brain injury, brain tumor)

Exclusion Criteria:

* Presence of hemispatial neglect (indexed by pathological asymmetries on paper-and-pencil tests)
* Disorders of conjugated eye movements
* Other neurological disorders (e.g., dementia)
* Exclusion criteria for brain stimulation (i.e., epilepsy or family history of epilepsy; implanted electrodes, stimulators, pacemakers, infusion pumps, or any implanted metal device; pregnancy)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Accuracy on the EF Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 4-month follow-ups
  Computerized visual search task. Participants have to search for the target letter "F" surrounded by distractors "E"s. Accuracy: the proportion of correct responses (range 0-1).
Change from baseline in Response Times (RTs) on the EF Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 4-month follow-ups
  Computerized visual search task. Participants have to search for the target letter "F" surrounded by distractors "E"s. RTs: median search times (seconds) of correct responses.
Change from baseline in Accuracy on the Triangle Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 4-month follow-ups
  Computerized visual search task. Participants have to report the number of triangles (targets) surrounded by square distractors. Accuracy: the proportion of correct responses (range 0-1).
Change from baseline in RTs on the Triangle Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 4-month follow-ups
  Computerized visual search task. Participants have to report the number of triangles (targets) surrounded by square distractors. RTs: median search times (seconds) of correct responses.
Change from baseline in RTs on the Numbers Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 4-month follow-ups
  Computerized visual search task. Participants have to point to numbers (1 to 15) in ascending order. RTs: median search times (seconds).
Change from baseline in the functional scale assessing the impact of vision loss in everyday life activities | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 4-month follow-ups
  A scale assessing the impact of HVFDs on nine activities of daily living. For each item, the score ranges from 0 ("No difficulty") to 4 ("Very frequent difficulties").

SECONDARY OUTCOMES:
Change from baseline in Accuracy on the Visual Detection Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 4-month follow-ups
  Detection of visual stimuli presented on the same panel employed for the training. Accuracy (the proportion of detected stimuli; range 0-1) is calculated for both the sighted and the blind hemifields.
Change from baseline in RTs on the Visual Detection Task | At baseline (at the beginning of the treatment), at the end of the treatment, at 1- and 4-month follow-ups
  Detection of visual stimuli presented on the same panel employed for the training. RTs: median search times of the detected stimuli are calculated for both the sighted and the blind hemifields.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual, anonymized, data will be uploaded on Zenodo.
Time Frame: Upon the publication of the study
Access Criteria: Access to data will be granted upon request

REFERENCES:
- [Background] Bolognini N, Rasi F, Coccia M, Ladavas E. Visual search improvement in hemianopic patients after audio-visual stimulation. Brain. 2005 Dec;128(Pt 12):2830-42. doi: 10.1093/brain/awh656. Epub 2005 Oct 11. PMID 16219672
- [Background] Bolognini N, Fregni F, Casati C, Olgiati E, Vallar G. Brain polarization of parietal cortex augments training-induced improvement of visual exploratory and attentional skills. Brain Res. 2010 Aug 19;1349:76-89. doi: 10.1016/j.brainres.2010.06.053. Epub 2010 Jul 1. PMID 20599813
- [Derived] Diana L, Casati C, Melzi L, Marzoli SB, Bolognini N. Enhancing multisensory rehabilitation of visual field defects with transcranial direct current stimulation: A randomized clinical trial. Eur J Neurol. 2025 Jan;32(1):e16559. doi: 10.1111/ene.16559. Epub 2024 Nov 28. PMID 39607286